CLINICAL TRIAL: NCT04295187
Title: Physical, Mental and Motor Development of Children Born to Mothers Treated With Pessary or Progesterone Supplement for Preventing Preterm Birth
Brief Title: Health of Pessary Versus Progesterone Supplement for Preventing Preterm Birth Children
Status: Completed | Type: Observational
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: CS/BVMĐ/20/03
Record Dates: First submitted 2020-03-02; First posted 2020-03-04 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Preterm Birth
Keywords: Pesary; Progesterone; ASQ-3; Health of children
MeSH Terms: conditions — Premature Birth | interventions — Health Status

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cervical pessary: Cervical pessary (Arabin) will be inserted to participants at 16-22 weeks and removed at 37 weeks of pregnancy or in case of premature rupture of membranes, signs of preterm labour or patient severe discomfort.
  Interventions: Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3; Other: Physical development and General Health; Other: Developmental Red flags
- Vaginal Progesterone: Vaginal progesterone (Cyclogest 200 mg) once a day will be used, from 16-22 to 37 weeks of pregnancy or in case of premature rupture of membranes, signs of preterm labour or patient severe discomfort.
  Interventions: Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3; Other: Physical development and General Health; Other: Developmental Red flags

INTERVENTIONS:
Other: Developmental score according to The Ages & Stages Questionnaires®, Third Edition - ASQ®-3 — Ages & Stages Questionnaires®, Third Edition (ASQ®-3) is a developmental screening tool designed for use by early educators and health care professionals. It relies on parents as experts, is easy-to-use, family-friendly and creates the snapshot needed to catch delays and celebrate milestones.
Other: Physical development and General Health — Physical development and General health examination
Other: Developmental Red flags — Developmental Red flags Questionnaires

SUMMARY:
To give strong recommendations on the efficacy and safety of vaginal progesterone versus cervical cerclage, we conduct this study to investigate the physical and mental development of children from vaginal progesterone versus cervical cerclage. Based on our research (Dang et al., 2019), the twin pregnancies with cervical lengths less than 38mm were randomly assigned to receive vaginal progesterone or cervical cerclage, which leads to the similarity in characteristics of these two groups. Hence, the result of analyzing these offsprings would be preciously valuable.

DETAILED DESCRIPTION:
Preterm birth (PB) is the leading cause of neonatal morbidity and mortality. Twin pregnancies and short cervical length are two high-risk factors of PB. Generally, in singleton pregnancies with short cervical length below 25 mm, or with a history of preterm birth, preventive measures of PB are vaginal progesterone and cervical cerclage. The cervical pessary is also being investigated for effectiveness in PB prevention in different populations. However, the effective preventive methods for PB has not been identified up to now in twin pregnancies with short cervical length.

In our research, the results showed that the preterm birth rate before 34 weeks in the cervical pessary group was lower than the progesterone group (16% vs 22%, RR 0.73; 95% CI 0.46 - 1.18). The perinatal outcomes were also better in the cervical pessary group than in the progesterone group (19% vs 27%, RR 0.70; 95% CI 0.43 - 0.93). The cost of the cervical pessary method was also significantly lower than the vaginal progesterone method cost. Pessary insertion was also more convenient since it was only inserted once during pregnancy, compared to daily vaginal progesterone. Therefore, the cervical pessary may be an appropriate option for preventing preterm birth in twin pregnancies with a short cervix.

However, besides these short-term outcomes, we need to pay more attention to the longer-term issues of both mothers and infants. Some evidence up to now has demonstrated that both these two methods are safe with no impact on physical, mental, and motor development of children up to 3 years old and even in older children. However, such evidence is still rare. Also, there hasn't been any study evaluating the impact, if any, of these two PB preventive methods.

ELIGIBILITY:
Inclusion Criteria:

* Live babies born from The pessary versus vaginal progesterone in women with a twin pregnancy and a cervix <38 mm study (NCT02623881)
* Parents agree to participate in the study.

Exclusion Criteria:

* Babies died after the perinatal period.

Ages: 1 Month to 66 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Live babies born following the pessary versus vaginal progesterone in women with a twin pregnancy and a cervix <38 mm study (NCT02623881)
Sampling Method: Non-Probability Sample
Enrollment: 529 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-12-09 (Actual)

PRIMARY OUTCOMES:
The average total ASQ-3 score | Up to 66 months after birth
  ASQ-3 (Ages and Stages Questionaires®) has 5 aspects: Communication, Gross motor, Fine motor, Problem solving and Personal-Social Each aspect has 6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0.
  ASQ-3 average = average score of 5 aspects.

SECONDARY OUTCOMES:
Score of Communication | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Gross motor | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Fine motor | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Problem solving | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
Score of Personal-Social | Up to 66 months after birth
  6 questions, if the answer is Yes, score = 10, Sometimes = 5 and Not yet = 0. Total score will be used: minimum = 0 and maximum = 60. Each aspects in each stages has alternative threshold
The rate of children who have at least one red flag sign | From 2 to 5.5 years after birth
  He or she has at least one red flag sign by age
  From 2 to < 3 year-old:
  Has very unclear speech Doesn't understand simple instruction • Doesn't speak in sentences Doesn't make eye contact Loses skills he/she once had
  From 3 to < 4 year-old:
  Can't jump in place Doesn't play pretend or make-believe • Speaks unclearly Can't retell a favorite story Doesn't use "me" and "you" correctly Loses skills he/she once had
  From 4 to < 5.5 year-old:
  Is easily distracted, has trouble focusing on one activity for more than 5 minutes • Doesn't talk about daily activities or experiences Shows extreme behavior Loses skills he/she once had
Duration of breast-feeding | Up to 24 months after birth
  Duration of breast-feeding
Infant age at which weaning starts | Up to 24 months after birth
  Infant age at which weaning starts
Name of diseases that lead to hospital admission | Up to 66 months after birth
  Name of diseases that lead to hospital admission
Number of hospital admission | Up to 66 months after birth
  Number of hospital admission
Weight | Through study completion, an average of 1.5 months
  Weight on the examination date
Height | Through study completion, an average of 1.5 months
  Height on the examination date

OTHER OUTCOMES:
The rate of long-term illness and chronic conditions | Up to 66 months after birth
  Any long-term illness and chronic condition appears in a child

CONTACTS AND LOCATIONS:
Overall Officials: Dang Q Vinh, MD, Principal Investigator — Mỹ Đức Hospital
Locations (1):
- Mỹ Đức Hospital, Ho Chi Minh City, Vietnam

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dang VQ, Nguyen LK, Pham TD, He YTN, Vu KN, Phan MTN, Le TQ, Le CH, Vuong LN, Mol BW. Pessary Compared With Vaginal Progesterone for the Prevention of Preterm Birth in Women With Twin Pregnancies and Cervical Length Less Than 38 mm: A Randomized Controlled Trial. Obstet Gynecol. 2019 Mar;133(3):459-467. doi: 10.1097/AOG.0000000000003136. PMID 30741812